CLINICAL TRIAL: NCT00690287
Title: A Dose-Ranging Study to Evaluate Fasting and Postprandial P-Glucose, Safety and Tolerability After Oral Single, B.I.D and Q.I.D Dosing of AZD6370 in Patients With Diabetes Mellitus: a Randomized, Single-Blind, Placebo-Controlled, Phase I Study
Brief Title: A Study to Evaluate P-Glucose, Safety and Tolerability After Oral Single Dosing of AZD6370 in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D0280C00014
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)-5-(4-(methylsulfonyl)phenoxy)benzamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A, arm 1 (Experimental): 1) 8 pats: AZD6370 increasing oral single doses a+b+c+placebo together with food
  Interventions: Drug: AZD6370
- Part A, arm 2 (Experimental): 1) 8 pats: AZD6370 increasing oral single doses a+b+c+placebo without food
  Interventions: Drug: AZD6370
- Part B, arm1, 2, and 3 (Experimental): 1. AZD6370 dose x mg o.d.
  2. dose x/2 mg b.i.d.
  3. dose x/4 mg q.i.d.
  Interventions: Drug: AZD6370
- Part B, arm 4 (Experimental): 4) Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6370 — Oral single doses a+b+c, o.d., suspension
  Arms: Part A, arm 1; Part A, arm 2
Drug: AZD6370 — Oral single dose, o.d., b.i.d. and q.i.d., suspension
  Arms: Part B, arm1, 2, and 3
Drug: Placebo — Placebo
  Arms: Part B, arm 4

SUMMARY:
The purpose of this study is to assess the effect of AZD6370 on blood sugar and to study safety and tolerability in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Treated with diet or metformin. Stable glycemic control indicated by no changed treatment within 3 months
* Diabetes Mellitus diagnosis <5 years

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the investigator, within two weeks before the first administration of the investigational product
* Clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic variables | Blood samples taken repeatedly during 24 hours on study day sessions

SECONDARY OUTCOMES:
Safety variables | Blood samples taken repeatedly during 24 hours on study day sessions
Pharmacokinetic variables | Blood samples taken repeatedly during 24 hours on study day sessions

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Prof., Study Director — AstraZeneca R&D Mölndal, SE-431 83 Mölndal, Sweden; Wolfgang Kühn, MD, Principal Investigator — Quintiles AB, Phase I Services, Strandbodgatan 1, SE-753 23 Uppsala, Sweden
Locations (3):
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Luleå
  - Research Site, Uppsala

REFERENCES:
- [Derived] Ericsson H, Sjoberg F, Heijer M, Dorani H, Johansson P, Wollbratt M, Norjavaara E. The glucokinase activator AZD6370 decreases fasting and postprandial glucose in type 2 diabetes mellitus patients with effects influenced by dosing regimen and food. Diabetes Res Clin Pract. 2012 Dec;98(3):436-44. doi: 10.1016/j.diabres.2012.09.025. Epub 2012 Sep 23. PMID 23010558